CLINICAL TRIAL: NCT03573674
Title: SujuKE - Improving Work Flow Through Cognitive Ergonomics. An Intervention Study
Brief Title: Improving Work Flow Through Cognitive Ergonomics. An Intervention Study
Acronym: SujuKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute of Occupational Health (Other)
Collaborators: Finnish Work Environment Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 117155; 117155 (Other Grant/Funding Number: The Finnish Work Environment Fund)
Record Dates: First submitted 2018-05-24; First posted 2018-06-29 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Ergonomics
Keywords: Working conditions,; cognitive load; disruptions; interruptions; information overload; Mental contrasting with implementation intentions MCII; Cognitive ergonomics

STUDY DESIGN:
Intervention Model Description: Cluster randomization with stratification allocated groups selected by participating organizations to treatment and control groups. Primary stratification was by the organization. Within-organization stratification took into account the size, the type of work tasks and the response rate in the first survey of cluster. Participating organizations entered all together to 36 clusters, each with individuals for the intervention and active control groups (N=638 individuals). The intervention (and active control) receive different types of workshops, individual tasks and team tasks. Additional information is available from non-randomized passive control group (N=289 individuals).
  Participating organizations were recruited by informing about the study. Participating units included knowledge workers, whose work tasks are cognitively rather than physically demanding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive ergonomics Intervention (Experimental)
  Interventions: Behavioral: CE - Cognitive Ergonomics (KERGO)
- Stress management Intervention (Active Comparator)
  Interventions: Behavioral: RS - Recovery Support (KUORMA)
- Passive control (No Intervention): "Passive Control" groups receive no intervention at all.

INTERVENTIONS:
Behavioral: CE - Cognitive Ergonomics (KERGO) — CE "Cognitive ergonomics Intervention" deals with themes such as disruptions, interruptions, information overload.
  A cognitive behaviour change method was applied in the intervention tasks. Both the tasks of discussing and developing new practices within the groups of individuals and the tasks for individuals were constructed to utilize mental contrasting with implementation intentions (MCII) method
  Arms: Cognitive ergonomics Intervention
Behavioral: RS - Recovery Support (KUORMA) — RS "Recovery Support / Stress Management Intervention" deals with themes such as workload management, recovery, work-family balance.
  A cognitive behaviour change method was applied in the intervention tasks. Both the tasks of discussing and developing new practices within the groups of individuals and the tasks for individuals were constructed to utilize mental contrasting with implementation intentions (MCII) method
  Arms: Stress management Intervention

SUMMARY:
The main aim of the SujuKE study is to test the effectiveness of workplace cognitive ergonomics development program designed to decrease cognitively disrupting work conditions and work-related cognitive stress, and to improve work flow. The cognitive ergonomics workplace intervention includes cognitive ergonomics workshop, work experiments, and intervention task questionnaires. Its effect on changes in subjective measures of work conditions, work flow, stress, and work productivity will be studied. The hypothesis is that cognitive ergonomics intervention decreases the level of cognitive strain related to work conditions, and this change is associated with higher level in work flow, well-being, and productivity at work.

DETAILED DESCRIPTION:
In the modern work life, performing work tasks rely on cognitive function, i.e. mental processes that are involved in processing information, such as attention, working memory, decision making and learning. Furthermore, the conditions at work include situations that require cognitive capacity. Information overload, multitasking and interruptions are typical features in any work. Thus, in the modern work life, work is knowledge work or information work by nature, and cognitive strain is a notable psychosocial risk factor. Not only task demands per se can exceed natural limitations of human cognitive capacities, but also the conditions at work can make it demanding for a human to perform.

Research shows that psychosocial stress, including cognitive stress, challenges wellbeing, safety and productivity at work. Cognitively straining conditions, such as disruptions, interruptions and information overload are related to higher levels of work stress, occupational accidents, and cognitive failures at work. It is essential to decrease harmful consequences to individual workers, organizations, and the society by managing psychosocial risks typical to cognitively demanding work tasks and conditions.

SujuKE study focuses on ergonomics (or human factors) practices that aim to ensure 'appropriate interaction between work, product and environment, and human needs, capabilities and limitations'. In cognitive ergonomics, the focus is on making human-system interaction compatible with human cognitive abilities and limitations, particularly at work. The aim is to apply general principles and good practices of cognitive ergonomics that help to avoid unnecessary cognitive load at work and that improve human performance.

The aim of the SujuKE study is to improve the conditions of knowledge work and promote the flow of work and reduce work strain. There are studies which show that decreasing disruptions, providing uninterrupted working time, and reducing information may lead to improved work flow and productivity. In the SujuKE-study, several sources of cognitive strain are restricted and concrete methods to help improve cognitive ergonomics will be worked on and implemented at workplace. The objective of the project is to obtain research evidence of the effects of cognitive ergonomics development programme on working conditions, the flow of work, well-being at work, and the productivity at work.

During the SujuKE project, the investigators will implement measures at the workplace that aim to facilitate work and reduce strain. The objective of the project is to obtain research evidence of the effects of these measures on working conditions, the flow of work, well-being at work, and the productivity at work. The study is carried out by the Finnish Institute of Occupational Health (FIOH) and funded by the Finnish Work Environment Fund.

ELIGIBILITY:
The participants in the study work in the participating organizations were recruited through direct contacts and by informing about the study in various events.

Inclusion Criteria:

* The participating organization offers several comparable teams (regarding type of tasks and demands) for study
* The participating units (in organizations) include knowledge workers, such as office workers and experts

Whose

* work tasks are cognitively rather than physically demanding
* work requires learning and updating knowledge and skills
* information and communication technology is the main tool at work.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 927 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Change in cognitive strain prevalence | 1: Baseline measurements: 10-16 weeks before the intervention phase. 2: End-of-treatment measurements: 18-28 weeks after the baseline measurements. 3: Follow-up 4m: 16 weeks after the end-of-treatment. 4: Follow-up 10m: 40 weeks after end-of-treatment
  Cognitive strain prevalence measures prevalence of disruptions, interruptions, and information overload.
  There are two items on disruptions, three items on interruptions, and seven items on information overload including memory load, multitasking, and problems with instructions (Brain@Work survey by FIOH).
  Response scale is from 1 to 5, higher number indicating higher prevalence (Scale: More rarely; Monthly; Weekly; Daily, or almost daily; Many times a day) Total score is a factor score including all 12 items.

SECONDARY OUTCOMES:
Change in subjective Cognitive load | 1: Baseline measurements: 10-16 weeks before the intervention phase. 2: End-of-treatment measurements: 18-28 weeks after the baseline measurements. 3: Follow-up 4m: 16 weeks after the end-of-treatment. 4: Follow-up 10m: 40 weeks after end-of-treatment
  Measured a) for the main themes of the intervention study. There are two items on disruptions, three items on interruptions, and seven items on information overload including memory load, multitasking, and problems with instructions (Brain@Work survey by FIOH).
  Furthermore, measured b) with all 39 items from FIOH Brain@Work Index questionnaire including 13 subscales.
  Response scale is from -3 to 3 (seven-point), negative values reflecting motivation-energization, positive values reflecting strain, zero reflecting neither. Higher number indicates higher load (Scale: Motivate-Energize Very much; Quite a lot; Somewhat; Cause strain Somewhat; Quite a lot; Very much).
  Total scores are averaged a) over the 12 items (disruptions, interruptions, information overload) and b) over the 39 items (all 13 subscales) weighted with their estimated prevalence (5 point scale, higher values reflecting higher prevalence).
Change in Recovery | 1: Baseline measurements: 10-16 weeks before the intervention phase. 2: End-of-treatment measurements: 18-28 weeks after the baseline measurements. 3: Follow-up 4m: 16 weeks after the end-of-treatment. 4: Follow-up 10m: 40 weeks after end-of-treatment
  Includes 1 item recovery measure. Measured with question: "How well do you usually feel that you recover from the strain caused by your work (both mental and physical) after your working day/work shift?". Scale from 0 (very poorly) to 10 (very well).
Change in stress | 1: Baseline measurements: 10-16 weeks before the intervention phase. 2: End-of-treatment measurements: 18-28 weeks after the baseline measurements. 3: Follow-up 4m: 16 weeks after the end-of-treatment. 4: Follow-up 10m: 40 weeks after end-of-treatment
  Includes 1 item stress measure. Measured with question "By stress we mean a situation in which a person feels tense, restless, nervous, or anxious, or they find it difficult to sleep because they cannot switch off their thoughts. Do you currently feel this kind of stress? (Choose the option that best suits you)". Scale from 0 (not at all) to 10 (very much).
Change in Burnout index | 1: Baseline measurements: 10-16 weeks before the intervention phase. 2: End-of-treatment measurements: 18-28 weeks after the baseline measurements. 3: Follow-up 4m: 16 weeks after the end-of-treatment. 4: Follow-up 10m: 40 weeks after end-of-treatment
  Burnout is measured with The Copenhagen Psychosocial Questionnaire II (COPSOQ-II) Burnout Index (Pejtersen, Kristensen, Borg, & Bjorner, 2010). The index includes four items. Scale: Not at all; A small part of the time; Part of the time; A large part of the time; All the time). Each item is scored 0-100 (0, 25, 50, 75, and 100), higher values indicating higher level of burnout. Total score is averaged over the four items.
Change in General health | 1: Baseline measurements: 10-16 weeks before the intervention phase. 2: End-of-treatment measurements: 18-28 weeks after the baseline measurements. 3: Follow-up 4m: 16 weeks after the end-of-treatment. 4: Follow-up 10m: 40 weeks after end-of-treatment
  Includes 1 item general health measure. Measured with question: "In general: would you say that your health is:" Scale: from 1 to 5, higher number indicating better health (Poor, Fairly poor, Average, Fairly good, Good).
Change in subjective presenteeism | 1: Baseline measurements: 10-16 weeks before the intervention phase. 2: End-of-treatment measurements: 18-28 weeks after the baseline measurements. 3: Follow-up 4m: 16 weeks after the end-of-treatment. 4: Follow-up 10m: 40 weeks after end-of-treatment
  Presenteeism / Subjective productivity Health at Work (HPQ) survey (World Health Organization, WHO 2001) questions B14: how would you rate your usual job performance over the past year or two? (Scale 0-10 with 10 being top performance) and B15: how would you rate your overall job performance on the days you worked during the past 4 weeks (28 days)? (Scale 0-10 with 10 being top performance)
Change in Cognitive stress symptoms | 1: Baseline measurements: 10-16 weeks before the intervention phase. 2: End of treatment measures: 18-28 weeks after baseline.
  Cognitive stress symptoms are measured with COPSOPQ-II Cognitive Stress Index (Pejtersen, Kristensen, Borg, & Bjorner, 2010). The index includes four items (scale: Not at all; A small part of the time; Part of the time; A large part of the time; All the time). Each item is scored 0-100 (0, 25, 50, 75, and 100), higher values indicating higher level of stress symptoms.
  Total score is averaged over the four items.
Change in Work flow | 1: Baseline measurements: 10-16 weeks before the intervention phase. 2: End of treatment measures: 18-28 weeks after baseline. .
  Work flow is measured as cognitive failure at work with three subscales. a) Workplace Cognitive Failure Scale (WCFS) memory sub-scale includes five items, b) WCFS attention sub-scale includes five items (Wallace & Chen 2005), and c) FIOH Cognitive failure: Multitasking subscale includes three items.
  The scale is from one to five (More rarely; Monthly; Weekly; Daily, or almost daily; Many times a day), higher number indicating higher prevalence of cognitive failure and lower work flow.
  Total scores are averaged for each subscale: WCFS memory, WCFS attention, and FIOH multitasking.

CONTACTS AND LOCATIONS:
Overall Officials: Virpi SS Kalakoski, Dr, Principal Investigator — Finnish Institute of Occupational Health
Locations (1):
- Finnish Institute of Occupational Health, Helsinki, Etelä-Suomi, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalakoski V, Selinheimo S, Valtonen T, Turunen J, Kapykangas S, Ylisassi H, Toivio P, Jarnefelt H, Hannonen H, Paajanen T. Effects of a cognitive ergonomics workplace intervention (CogErg) on cognitive strain and well-being: a cluster-randomized controlled trial. A study protocol. BMC Psychol. 2020 Jan 2;8(1):1. doi: 10.1186/s40359-019-0349-1. PMID 31898551